CLINICAL TRIAL: NCT01654874
Title: 99mTc-MIP-1404 for Imaging Prostate Cancer: Phase I Clinical Study to Assess the Image Quality of a Simplified Kit Formulation Compared to a Multi-step Preparation of 99mTc-MIP-1404
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: MIP-TcTx-P101b
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — technetium 99m 1-(1-(2-(bis(carboxymethyl)amino)-2-oxoethyl)-1H-imidazol-2-yl)-2-((1-(2-(bis(carboxymethyl)amino)-2-oxoethyl)-1H-imidazol-2-yl)methyl)-9,14-dioxo-2,8,13,15-tetraazaoctadecane-7,12,16,18-tetracarboxylic acid)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preparation A (Experimental): 20 (±3) mCi 99mTc-MIP-1404 (preparation A)
  Interventions: Drug: 99mTc-MIP-1404
- Preparation B (Experimental): 20 (±3) mCi 99mTc-MIP-1404 (preparation B)
  Interventions: Drug: 99mTc-MIP-1404

INTERVENTIONS:
Drug: 99mTc-MIP-1404

SUMMARY:
This trial is a single-blind, cross-over design. Up to three patients with confirmed metastatic prostate adenocarcinoma and up to three healthy volunteers will receive two doses of 20.0 (± 3) mCi of intravenously administered 99mTc MIP 1404 (preparation A or preparation B). Whole-body planar scintigraphic images will be acquired at various time points on the day of study drug administration. A pelvic SPECT/CT image will be acquired on the day of study drug administration. Blood will be collected for pharmacokinetic measurements following study drug administration. Each participant will receive an initial study drug administration (preparation A) and a second study drug administration (preparation B) approximately 7 to 21 days later. A final follow-up visit will occur approximately 2 - 3 weeks after the second study drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 21 years or older.
* Ability to provide signed informed consent and willingness to comply with protocol requirements.
* Participants must agree to use an acceptable form of birth control throughout the study period. Participants must agree to use condoms for a period of seven days after each study drug administration, if engaged in sexual activity.

Additional Inclusion Criteria for Metastatic Prostate Adenocarcinoma Patients:

* Histologic diagnosis of prostate cancer by validated medical history (pathology report, if available).
* Evidence of metastatic disease demonstrated by a documented abnormal bone scan, CT scan, or MRI
* Karnofsky performance is ≥ 60

Additional Inclusion Criteria for Healthy Volunteers:

* PSA laboratory assessment within normal range (PSA < 4 ng/ml)
* Normal findings on a digital rectal examination
* Hemoglobin and hematocrit within normal range

Exclusion Criteria:

* Received a radioisotope within 5 physical half lives of that radioisotope prior to study enrollment
* Have any medical condition or other circumstances which, in the opinion of the Investigator, would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or post dose follow-up examinations
* Participant is determined by the Investigator to be clinically unsuitable for the study
* Serum creatinine ≥ 2.0 mg/dl
* Total bilirubin ≥ 2.0 mg/dl
* Liver transaminases ≥ 1.5 x ULN
* Platelet count < 100,000/mm3
* Absolute neutrophil count (ANC) < 2,000/mm3
* Hematocrit < 30% or hemoglobin < 10 g/dl

Additional Exclusion Criteria for Metastatic Prostate Adenocarcinoma Patients:

* Have received a permanent prostate brachytherapy implant within the last 3 months for 103Pd implants; or 12 months for 125I implants
* Have had any other malignancies within the past year, other than basal or squamous cell carcinoma of the skin, in which the diagnosis and location have not been defined as clinically controlled or treated to complete response

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To assess the image quality of a simplified kit formulation of 99mTc-MIP-1404 (study drug) compared to a multi-step preparation of 99mTc-MIP-1404 in patients with confirmed metastatic prostate adenocarcinoma and in healthy volunteers | Whole-body planar scintigraphic images will be acquired at 30 min, 2 and 4 hours post administration. A pelvic SPECT/CT image will be acquired at 3 hours post study drug administration

SECONDARY OUTCOMES:
To determine the pharmacokinetics, biodistribution and tumor uptake of 99mTc-MIP-1404 preparations in patients with confirmed metastatic prostate adenocarcinoma and in healthy volunteers | Blood will be collected for PK and radioactivity counting at baseline, 2 minutes, 5 minutes, 30 minutes, 1 hour, 2 hours, and 4 hours post study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley J Goldsmith, MD, Principal Investigator — Department of Nuclear Medicine, New York Presbyterian Hospital, Weill Cornell Medical College
Locations (1):
- New York Presbyterian Hospital, Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Background] Pinto JT, Suffoletto BP, Berzin TM, Qiao CH, Lin S, Tong WP, May F, Mukherjee B, Heston WD. Prostate-specific membrane antigen: a novel folate hydrolase in human prostatic carcinoma cells. Clin Cancer Res. 1996 Sep;2(9):1445-51. PMID 9816319
- [Background] Smith-Jones PM, Vallabahajosula S, Goldsmith SJ, Navarro V, Hunter CJ, Bastidas D, Bander NH. In vitro characterization of radiolabeled monoclonal antibodies specific for the extracellular domain of prostate-specific membrane antigen. Cancer Res. 2000 Sep 15;60(18):5237-43. PMID 11016653
- [Background] Ghosh A, Heston WD. Tumor target prostate specific membrane antigen (PSMA) and its regulation in prostate cancer. J Cell Biochem. 2004 Feb 15;91(3):528-39. doi: 10.1002/jcb.10661. PMID 14755683
- [Background] Kinoshita Y, Kuratsukuri K, Landas S, Imaida K, Rovito PM Jr, Wang CY, Haas GP. Expression of prostate-specific membrane antigen in normal and malignant human tissues. World J Surg. 2006 Apr;30(4):628-36. doi: 10.1007/s00268-005-0544-5. PMID 16555021
- [Background] Murphy GP, Elgamal AA, Su SL, Bostwick DG, Holmes EH. Current evaluation of the tissue localization and diagnostic utility of prostate specific membrane antigen. Cancer. 1998 Dec 1;83(11):2259-69. PMID 9840525
- [Background] Vallabhajosula S, Kuji I, Hamacher KA, Konishi S, Kostakoglu L, Kothari PA, Milowski MI, Nanus DM, Bander NH, Goldsmith SJ. Pharmacokinetics and biodistribution of 111In- and 177Lu-labeled J591 antibody specific for prostate-specific membrane antigen: prediction of 90Y-J591 radiation dosimetry based on 111In or 177Lu? J Nucl Med. 2005 Apr;46(4):634-41. PMID 15809486
- [Background] Olson WC, Heston WD, Rajasekaran AK. Clinical trials of cancer therapies targeting prostate-specific membrane antigen. Rev Recent Clin Trials. 2007 Sep;2(3):182-90. doi: 10.2174/157488707781662724. PMID 18474004
- [Background] Rajasekaran AK, Anilkumar G, Christiansen JJ. Is prostate-specific membrane antigen a multifunctional protein? Am J Physiol Cell Physiol. 2005 May;288(5):C975-81. doi: 10.1152/ajpcell.00506.2004. PMID 15840561
- [Background] Slovin SF. Targeting novel antigens for prostate cancer treatment: focus on prostate-specific membrane antigen. Expert Opin Ther Targets. 2005 Jun;9(3):561-70. doi: 10.1517/14728222.9.3.561. PMID 15948673
- [Background] Wang X, Yin L, Rao P, Stein R, Harsch KM, Lee Z, Heston WD. Targeted treatment of prostate cancer. J Cell Biochem. 2007 Oct 15;102(3):571-9. doi: 10.1002/jcb.21491. PMID 17685433
- [Background] Barrett PH, Bell BM, Cobelli C, Golde H, Schumitzky A, Vicini P, Foster DM. SAAM II: Simulation, Analysis, and Modeling Software for tracer and pharmacokinetic studies. Metabolism. 1998 Apr;47(4):484-92. doi: 10.1016/s0026-0495(98)90064-6. PMID 9550550
- [Background] Stabin MG, Siegel JA. Physical models and dose factors for use in internal dose assessment. Health Phys. 2003 Sep;85(3):294-310. doi: 10.1097/00004032-200309000-00006. PMID 12938720
- [Background] Stabin MG, Sparks RB, Crowe E. OLINDA/EXM: the second-generation personal computer software for internal dose assessment in nuclear medicine. J Nucl Med. 2005 Jun;46(6):1023-7. PMID 15937315
- [Background] Pan ZY, Wolf W. Computer package for the calculation of the radiation dose to patients, based on the MIRD approach. J Nucl Med. 1985 Mar;26(3):318-20. No abstract available. PMID 3882906